CLINICAL TRIAL: NCT02722252
Title: Comparative Study of Two Embryo Culture Systems: Randomization of Attempts at In Vitro Fertilization With ICSI at the Centre for Medically Assisted Procreation at Dijon CHU
Brief Title: Comparative Study of Two Embryo Culture Systems
Acronym: INCUBATE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: FAUQUE - INCUBATE
Record Dates: First submitted 2016-03-18; First posted 2016-03-29 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Infertility
Keywords: In Vitro Fertilization with ICSI
MeSH Terms: conditions — Infertility | interventions — Fetoscopes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Embryoscope group
  Interventions: Device: Embryoscope
- Embryo culture without incorporated camera group
  Interventions: Device: Embryo culture system without incorporated camera

INTERVENTIONS:
Device: Embryoscope
  Groups: Embryoscope group
Device: Embryo culture system without incorporated camera
  Groups: Embryo culture without incorporated camera group

SUMMARY:
The centre for Medically-Assisted Procreation (MAP) of Dijon CHU has two high-technology embryo culture systems, with incubation characteristics that are potentially superior to those provided by classical culture systems. Indeed, these two systems, available in only two MAP centres in France, make it possible to maintain a stable temperature and gaseous environment during the in-vitro development of the embryos.

It is necessary to observe the development of the embryos to determine which embryos have the highest implantation potential. These observations are done from time to time by microscope for one system and continuously using an incorporated video camera for the other (cinematographic study). The MAP centre in Dijon wishes to compare the interest of these two systems.

ELIGIBILITY:
Inclusion Criteria:

* Persons who have provided oral consent
* Attempt at In Vitro Fertilization with ICSI (IntraCytoplasmic Sperm Injection)
* At least 6 mature ovocytes to microinject

Exclusion Criteria:

* Persons not covered by national health insurance
* Attempt at In Vitro Fertilization (IVF)
* Fewer than 6 mature ovocytes
* Decision to transfer at the zygote stage during the multidisciplinary meeting
* Attempts made in a context of viral risk (both systems are in a virus risk-free zone)
* Attempts with surgically-harvested spermatozoa

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Couples who attempt In Vitro Fertilization with ICSI (IntraCytoplasmic Sperm Injection)
Sampling Method: Probability Sample
Enrollment: 388 (Actual)
Dates: Start 2014-08-27 (Actual); Primary Completion 2017-03-29 (Actual); Study Completion 2017-03-29 (Actual)

PRIMARY OUTCOMES:
Implantation rate | 16 weeks after transfer
  The implantation rate is defined as the number of embryos implanted (gestational sacs seen on the US scan) compared to the total number of embryos transferred.

SECONDARY OUTCOMES:
Rate of miscarriages | 16 weeks after transfer

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de DIJON, Dijon, France

REFERENCES:
- [Result] Barberet J, Chammas J, Bruno C, Valot E, Vuillemin C, Jonval L, Choux C, Sagot P, Soudry A, Fauque P. Randomized controlled trial comparing embryo culture in two incubator systems: G185 K-System versus EmbryoScope. Fertil Steril. 2018 Feb;109(2):302-309.e1. doi: 10.1016/j.fertnstert.2017.10.008. Epub 2017 Nov 23. PMID 29175066